CLINICAL TRIAL: NCT02217137
Title: Analysing Tear Protein, Conjunctival Cells, and Imaging Eyes in Patients With Rheumatoid Arthritis and Systemic Lupus Erythematosus
Brief Title: Tear Proteins, Conjunctival Cells and Imaging Eyes in Rheumatoid Arthritis and Systemic Lupus Erythematosus Patients
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Other Study IDs: R1108/10/2014; 2014/269/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2014-06-09; First posted 2014-08-15 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-06

CONDITIONS: Dry Eye
Keywords: Dry Eye; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Tear cytokines and immune response
MeSH Terms: conditions — Dry Eye Syndromes; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Tear samples will be collected from the schimers strips for protein analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
Rheumatoid Arthritis (RA) and Systemic Lupus Erythematosus (SLE) are chronic systemic autoimmune diseases that have been reported to affect the ocular surface of patients [1,2]. However, the nature of the disturbances of the ocular surface immunity and their relationship to systemic disease severity are poorly understood.

This study aims to profile the ocular surface inflammation of RA and SLE patients by a., analysing levels of tear cytokine, and b., investigating conjunctival cells, and c. clinical imaging for conjunctival redness and tear stability.

20 consecutive RA patients and 20 consecutive SLE patients will be recruited from the Singapore General Hospital Rheumatology clinic. 20 age matched controls for SLE and another 20 age matched controls for RA will be recruited.

All participants will undergo

1. Tear collection with Schirmer strips
2. EyePRIMTM (Opia Technologies) Impression Cytology Device for conjunctival sampling
3. Clinical ocular surface assessment with Oculus Keratograph 5M
4. Collection of blood via venipuncture (optional)
5. Retrieval of Clinical Information of participants

The association of cytokines in the tears with various cellular and immune markers, as well as clinical signs of inflammation and tear stability will be investigated. This will be useful for further longitudinal studies of treatment in autoimmmune disease patients.

DETAILED DESCRIPTION:
Background and Rationale

Inflammatory autoimmune disease and eye involvement Rheumatoid Arthritis (RA) and Systemic Lupus Erythematosus (SLE) are chronic systemic autoimmune diseases of unknown etiology [2]. Ocular manifestations may range from conditions which cause distressing symptoms of discomfort, such as dry eye syndrome, to potentially sight-threatening conditions such as retinal vasculitis. The ocular surface is agreed to be the site most commonly affected by systemic autoimmune diseases, manifesting as dry eye syndrome. However, its related complications are poorly addressed [1,2]. The severity of ocular surface inflammation may be related to systemic immunology since systemic treatment will alter the signs of ocular surface disease.

EyePRIMTM (Opia Technologies) Impression Cytology Device Studies have shown that this method of combining flow cytometry with OSIC is useful to phenotype recovered cells from the superficial layers of the ocular surface [3]. There has been recent advances in clinical techniques for obtaining conjunctival cells for reseach studies. An example of an award winning device is the EyePRIMTM (Opia Technologies).

Previous studies have shown that EyePRIMTM is able to obtain sufficient cells for flow cytometry for immune markers [4]. In the study, the ocular surface of three healthy patients were analysed using EyePRIMTM and conventional semi-circular Supor PES filters for flow cytometry. One EyePRIMTM was used to impression the lateral bulbar conjunctiva and a second, the medial bulbar conjunctiva of the same eye. Cells were recovered from both EyePRIMTM using gentle agitation with a pipette tip for one minute, and then stained with antibody markers for leukocytes (CD45), CD16, epCAM, HLA-DR and a dead cell exclusion dye. Results have shown that the mean corrected total cell count collected using EyePRIMTM was greater than conventional methods (475,544 cells vs 335,226 cells). Out of the total cells collected, the mean corrected number of lymphocytes found via staining with CD45 antibody was around 1000.

Advances in clinical phenotyping Dry eye is a common ocular surface disease mediated by inflammation. It is postulated that dry eye in the context of systemic autoimmune diseases is caused by the infiltration of activated T lymphocytes into the bulbar conjunctiva, beginning a vicious cycle of chronic inflammation of the ocular surface [5]. In the dry eye database at SNEC/SERI (unpublished data), we found higher levels of fluorescein corneal staining, indicating presence of punctate epithelial erosions in patients with RA compared to dry eye patients without systemic autoimmune diseases. While we have not personally conducted studies on SLE patients, it is documented in existing literature that significant signs of dry eye have been detected in SLE patients using older assessment modalities such as the Schirmer's test and Rose Bengal staining [6].

Lastly, the availability of new phenotyping equipment such as the Oculus Keratograph 5M provides the opportunity for clinical parameters such as conjunctival redness and non-invasive tear break up time (NIBUT) to be assessed objectively, accurately and non-invasively [7]. To the best of the investigators' knowledge, these standardised tools have not been used in the context of rheumatological disease or its effect on the ocular surface.

Research experience at SERI In SERI there is significant experience with clinical and imaging studies of the ocular surface. The clinical profile of the ocular surface inflammation can be objectively measured or documented using newly available imaging techniques as described. In addition, a TCR grant will be jointly applied for in the coming months to examine systemic as well as ocular immune events during treatment of rheumatology patients including RA and SLE.

Preliminary data Our research team has experience with extraction of tear proteins from schirmer strips in a longitudinal trial and analysing after each patient's visit, tear cytokine concentrations for IL-1b, IL-2, IL-4, IL-6, IL-8, IL-10, IFN , TNFa , IL-12, IL-13, IL-17a, MCP, MIP1a, MMP9, IP10, RANTES using the BioPlex technique (Figure 1).

In other studies (unpublished data), our research group has successfully performed flow cytometry, and evaluated the proportion of various immune cell types by staining for cell surface markers. This study was performed on pterygium tissues. We were able to perform intracytoplasmic staining for cytokines after Phorbol Myristate Acetate (PMA) stimulation. This was performed for Th1 (eg. TNFα and IFN γ) and Th17 (eg. IL-17a) cytokines, from populations of T lymphocytes as few as 300-500.

1. HYPOTHESIS AND OBJECTIVES

Hypothesis and specific aims This study thus aims to profile the ocular surface inflammation of RA and SLE patients by a., analysing levels of tear cytokine, and b., investigating conjunctival cells, and c. clinical imaging for conjunctival redness and tear stability. In the conjunctiva of the patients, we expect to find conjunctival epithelial cells, stromal fibroblasts as well as various immune cells.

Study Objectives and Purpose

1. A primary purpose of the study is to profile A. tear cytokine levels and B. the proportion of various immune cells (eg., lymphocyte, dendritic cell and neutrophil subsets) in the conjunctival impressions.
2. The secondary aim is to further profile the immune response, either by examining the possible Th1 and Th17 responses of T cells to stimulation, or by the levels of inflammatory gene transcripts, ie., pattern of immune gene expression.
3. A third aim is to study the correlation between the activity of systemic disease, ocular surface status, and tear cytokine and immune cell levels of RA and SLE patients.

Outcomes 1. Tear cytokine levels 2. Conjunctival immune cell profile

1. Proportion of T lymphocytes and other immune cells
2. Immune gene expression 3. Clinical parameters for ocular surface: Conjunctival redness, tear meniscus height and NIBUT 4. Rheumatological disease activity indices of the patients

   Primary outcome:

   Tear cytokine levels and conjunctival immune cell profile of RA and SLE patients in comparison to healthy controls

   2. EXPECTED RIKS AND BENEFITS Expected risks No potential problems are expected for this study.

   Potential benefits With greater understanding of the presence of various inflammatory mediators, we can gain further insight into the complex process taking place. It is also possible that some markers like tear proteins can be biomarkers that warn individuals of systemic flares. We have jointly filed a provisional patent on such tear biomarkers in SLE flares. (Date of Filing: 11 September 2013 Singapore Provisional Patent Application No.: 201306892-9).

   3. STUDY POPULATION 3.1. List the number and nature of subjects to be enrolled. Participants and target sample size 20 consecutive RA patients and 20 consecutive SLE patients, aged 21 to 99, will be recruited from the Singapore General Hospital, under three settings a., SGH Rheumatology outpatients b., Rheumatology patients from the wards, c., Patients from pilot project under Dr Tan (CIRB REF: 2013/152/E).

   Permission would be sought from the attending doctors before subjects are being recruited. Eligible subjects will be counselled on the study by the study coordinator. If the subject is interested, the study coordinator will then accompany the subject to SERI for the relevant assessments. Informed written consent will be obtained from all participants.

   In addition, we will recruit 20 age matched controls for SLE and similarly another 20 controls for RA. If older controls are required, they will be from the pre-cataract patients, and younger ones from volunteers and other students. They will undergo the same assessments as the patients in the other groups. Publicity for the study will be carried out via posters or word of mouth (draft of poster is submitted for approval).

   3.2. Inclusion Criteria

   1. Clinically diagnosed with Rheumatoid Arthritis or Systemic Lupus Erythematosus.

   3.3. Exclusion Criteria

   All subjects meeting any of the exclusion criteria at baseline will be excluded from participation.

   1. Known history of thyroid disorders (diagnosed by physician). 2. No ocular surgery within the last 3 months and LASIK within 1 year. 3. Ocular surface diseases such as pterygium, or obvious lid/orbital disease with lagophthalmos.

   4. Any other specified reason as determined by clinical investigator.

   4. STUDY DESIGN AND PROCEDURES/METHODOLOGY

   Study Design:

   Prospective study

   No. of visits:

   There will only be 1 study visit in this study.

   Duration of Study:

   11 months (Apr 2014 to Mar 2015). Recruitment of patients and collection of data will take place from 22nd May 2014 to 31 July 2014.

   Procedures:

   The different procedures proposed in this small study are summarized below, and elaborated upon in subsequent paragraphs:
   1. Tear collection with Schirmer strips
   2. EyePRIMTM (Opia Technologies) Impression Cytology Device for conjunctival sampling
   3. Clinical ocular surface assessment with Oculus Keratograph 5M
   4. Collection of blood via venipuncture (optional)
   5. Retrieval of Clinical Information of participants

   <!-- -->

   1. a. Schirmer's I test This will be done with the standard strips currently used at SERI (5 mm wide with a notch for folding) (Schirmer Tear Test Strips, Clement Clarke International, UK). No prior anaesthetic will be used. The strips will be positioned over the temporal half of the lower lid margin in both eyes at the same time.

   The study participant will be asked to close their eyes. Any excessive irritation signs will be noted. The extent of the wetting in each strip will be recorded after 5 minutes of testing. The strip will be collected and stored in 1.5ml Eppendorf tubes at -80˚C until further cytokine analysis.

   1b. Tear cytokine level measurement with BioPlex Human Cytokine Assay We propose analyzing tear cytokine levels from tears collected on Schirmer strips. In previous studies on dry eye patients being treated with punctal occlusion, we were able to elute proteins from Schirmer strips and determine levels of 15 cytokines. Tear proteins will be extracted as in previous protocols at SERI [8]. Briefly, we will cut out the wetted portions of the strips and vortex after adding phosphate buffered saline in protease inhibitor.

   The assay will be using a commercially available bead based indirect sandwich immunofluorescence assay (Beadlyte Kit). The readout will be performed with the Bioplex (BIO-RAD) platform. Cytokine standard provided with the kit will be used to plot standard curves. The levels of cytokines in tears are normalised to per mm of Schirmer and further analysed. We believe this same method of tear-sample collection will be just as effective in assessing patients with RA/SLE.

   2. Impression cytology Impression cytology will be performed to collect the superficial conjunctiva cells for analysis. Conjunctiva impression specimen of the upper bulbar conjunctiva will be collected with the EyePRIMTM device.

   One drop of topical anaesthesia (eg. alcaine) is instilled. The eyelid will be held open with the thumb and forefinger. The distal end of the device will be positioned on the conjunctiva of the participant. The inner radius can be positioned adjacent to the limbus. The push-button will be pressed until the membrane is in contact with the temporal bulbar conjunctiva, holding for 2 to 3 seconds. It will then be removed from the conjunctiva with a peeling motion after 2-3 seconds. The membrane will subsequently be placed in RPMI 1640 medium supplemented with 10% heat-inactivated fetal calf serum.. This will be carried out over the temporal bulbar conjunctiva of both eyes. Each participant will then be given a single-use container of Refresh Plus ® artificial tears for self-application in case any ocular irritation is felt after impression cytology.

   The cells can then be processed after the patient's visit. Cells will be recovered from the EyePRIMTM filters using gentle agitation with a pipette tip for one minute, and then stained with antibody markers for dendritic cells (lymphoid and myeloid), NK cells, B cells, T cells , neutrophils and monocytes. Specifically, CD123, CD16, CD45, CD56, CD3, CD4, CD8, CD66b, CD11b, CD11c markers will be used.

   Cells harvested from impression cytology will be counted and undergo flow cytometry and depending on numbers, determination of the proportion of immune cells of various types, and even staining for Intracytoplasmic cytokines in lymphocytes after Phorbol Myristate Acetate stimulation. One modification of flow cytometry is the Amnis or microscopy coupled flow cytometry which can be performed at the SingHealth Immunology and Inflammation center. Amnis and microscopy couples flow cytometry can handle even less cells than conventional flow cytometry. If the cells from impression cytology are not sufficient for these purposes, nano-string transcript levels of various immune markers will be performed instead.

   3. Oculus K 5M imaging

a. Non-Invasive Tear Break-Up Time (Oculus K5M) Non-Invasive Tear Break-Up Time is measured non-invasively and fully automatically using Oculus K5M. The new infrared illumination is not visible to the human eye. This prevents glare during the examination. Patient will sit comfortably in front of the instrument and blink freely while fixing on a target directly ahead. Once the participant is ready, they will be instructed to blink twice and refrain from blinking. Keratograph 5M is fully automated and it will capture any break or distortion in the image and the time of the break will be noted. Three readings will be taken for each eye to get the average value.

b. Tear Meniscus Height (Oculus K5M) This can be measured non-invasively by the Oculus K5M to the nearest mm. Patient will sit comfortably in front of the instrument while fixing on a target directly ahead. Tear meniscus will be captured by the machine and tear meniscus height measured.

c. Conjunctival redness (Oculus K5M) Conjunctival redness will be assessed using Oculus K5M. Patient will sit comfortably in front of the instrument while fixing on a target directly ahead. Imaged will be captured and an overview display of conjunctival redness will be evaluated by "JENVIS Grading Scale".

4. Collection of blood via venipuncture (optional) 5-10ml of blood will be collected from patients via venipuncture. This is optional based on participant preference. Two different Participant Information Sheets have been prepared based on their choice of having venipuncture and disclosing its results. This will be taken on a non-study visit or when it is concurrent with a clinically indicated blood test.

5. Retrieval of Clinical Information of participants

Three areas of clinical information of the rheumatic status in our participants will be collected retrospectively. These areas are:

1. Most recent serology results for autoantibody titres and other blood test results such as erythrocyte sedimentation rate
2. History of drug prescriptions
3. Disease activity index and other relevant clinical information

We propose obtaining the data in 1) and 2) from the patient's electronic medical records via the Citrix XenApp portal. Disease activity index and other clinical information may be obtained from the case files of the patients.

Rationale Small volumes of fluid can be used in a multiplex way to determine more than one cytokine in the Beadlyte assay, compared to ELISA.

The EyePRIMTM technique is used because of prior studies that showed a high cellular yield and success in immune profiling with 3 healthy people.

Expected findings:

1. RA and SLE patients should have elevated tear cytokine levels and increased inflammatory cell population in their conjunctival samples.
2. RA and SLE patients should have greater signs of ocular surface inflammation than the healthy controls
3. The signs of ocular surface inflammation should correlate with disease activity, tear cytokines profiles and conjunctival inflammatory cell profiles.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Rheumatoid Arthritis or Systemic Lupus Erythematosus

Exclusion Criteria:

* Known history of thyroid disorders (diagnosed by physician).
* No ocular surgery within the last 3 months and LASIK within 1 year.
* Ocular surface diseases such as pterygium, or obvious lid/orbital disease with lagophthalmos.
* Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthriris, Systemic Lupus Erythematosus and healthy normal volunteers will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Profile tear cytokines | 1 day
  the inflammatory cytokines concentration

SECONDARY OUTCOMES:
Profile immune response | 1 day
  the levels of inflammatory gene transcripts, ie., pattern of immune gene expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore